CLINICAL TRIAL: NCT00682734
Title: Metoclopramide for Acute Migraine: A Dose Finding Study
Brief Title: Metoclopramide for Migraine: A Dose Finding Study
Acronym: MDFS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-11-405
Record Dates: First submitted 2008-05-19; First posted 2008-05-22 (Estimated); Results first posted 2012-12-31 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Metoclopramide; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Metoclopramide 10 mg+ diphenhydramine 25 mg. This medication was administered as an intravenous drip over 20 minutes
  Interventions: Drug: metoclopramide; Drug: Diphenhydramine 25mg
- 2 (Experimental): metoclopramide 20 mg + diphenhydramine 25 mg. Administered as an intravenous drip over 20 minutes.
  Interventions: Drug: metoclopramide; Drug: Diphenhydramine 25mg
- 3 (Experimental): metoclopramide 40 mg + diphenhdyramine 25mg. Administered as an intravenous drip over 20 minutes.
  Interventions: Drug: metoclopramide; Drug: Diphenhydramine 25mg

INTERVENTIONS:
Drug: metoclopramide — metoclopramide 20 mg
  Arms: 2
Drug: metoclopramide — metoclopramide 40 mg
  Arms: 3
Drug: metoclopramide — metoclopramide 10 mg
  Arms: 1
Drug: Diphenhydramine 25mg — Diphenhydramine 25mg, administered as an intravenous drip over 20 minutes

SUMMARY:
Metoclopramide is an effective intravenous treatment for acute migraine attacks, but we do not know the best dose to administer. This study compares three different doses of metoclorpamide.

DETAILED DESCRIPTION:
Patients with acute migraine attacks are eligible for enrollment if they present to the emergency department of Montefiore Medical Center. Pain scores are assessed at baseline and every 30 minutes for two hours, and then again by telephone 48 hours after discharge

ELIGIBILITY:
Inclusion Criteria:

* acute migraine

Exclusion Criteria:

* secondary cause of headache
* lumbar puncture
* allergy or intolerance to study medication

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W. Friedman, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metoclopramide 10 mg Intravenous: Metoclopramide 10 mg intravenous + diphenhydramine 25mg intravenous
- Metoclopramide 20 mg Intravenous: Metoclopramide 20 mg intravenous+ diphenhydrmaine 25 mg intravenous
- Metoclopramide 40 mg Intravenous: Metoclopramide 40 mg intravenous + diphenhdyramine 25 mg intravenous
Period: Emergency Department Portion
Arm/Group | Metoclopramide 10 mg Intravenous | Metoclopramide 20 mg Intravenous | Metoclopramide 40 mg Intravenous
Started | 113 | 118 | 118
Completed | 113 | 117 | 117
Not Completed | 0 | 1 | 1
Period: 48 Hour Follow-up
Arm/Group | Metoclopramide 10 mg Intravenous | Metoclopramide 20 mg Intravenous | Metoclopramide 40 mg Intravenous
Started | 113 | 117 | 117
Completed | 107 | 111 | 106
Not Completed | 6 | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Metoclopramide 10 mg Intravenous: Metoclopramide 10 mg intravenous + diphenhydramine 25 mg intravenous
- Metoclopramide 20 mg: Metoclopramide 20mg intravenous+ diphenhydrmaine 25 mg intravenous
- Metoclopramide 40 mg: Metoclopramide 40 mg intravenous + diphenhdyramine 25 mg intravenous
- Total: Total of all reporting groups
Arm/Group | Metoclopramide 10 mg Intravenous | Metoclopramide 20 mg | Metoclopramide 40 mg | Total
Number analyzed (Participants) | 113 | 118 | 118 | 349
Age, Continuous [Mean (Standard Deviation); unit: years]
  Adults | 38.7 (11.5) | 37.5 (9.9) | 38.4 (12.0) | 38.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 103 | 97 | 294
  Male | 19 | 15 | 21 | 55

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score
Description: Change in 11 point pain intensity score between baseline and one hour. At both baseline and one hour, all patients were asked to describe their pain on a scale from 0 to 10, with 0 signifying no pain and 10 signifying the worst pain imaginable. Therefore, the CHANGE in pain score could range from -10 through 10.
Time Frame: Baseline, 60 minutes
Population: per protocol
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Metoclopramide 10 mg Intravenous: Metoclopramide 10mg intravenous + diphenhydramine 25mg intravenous
- Metoclopramide 20 mg: Metoclopramide 20 mg intravenous+ diphenhydrmaine 25 mg intravenous
- Metoclopramide 40 mg: Metoclopramide 40mg intravenous + diphenhdyramine 25mg intravenous
Arm/Group | Metoclopramide 10 mg Intravenous | Metoclopramide 20 mg | Metoclopramide 40 mg
Number analyzed (Participants) | 113 | 117 | 117
scores on a scale | 4.7 (2.6) | 4.9 (2.8) | 5.3 (2.8)

ADVERSE EVENTS:
Arm/Group | Metoclopramide 10 mg Intravenous | Metoclopramide 20 mg | Metoclopramide 40 mg
Serious Adverse Events (participants affected / at risk) | 0/113 | 1/118 | 0/118
Other Adverse Events (participants affected / at risk) | 8/113 | 8/118 | 7/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide 10 mg Intravenous (N=113) | Metoclopramide 20 mg (N=118) | Metoclopramide 40 mg (N=118)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metoclopramide 10 mg Intravenous (N=113) | Metoclopramide 20 mg (N=118) | Metoclopramide 40 mg (N=118)
Akathisia (Nervous system disorders) | 8 | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes